CLINICAL TRIAL: NCT05627375
Title: Best Antithrombotic Therapy in Patients With Acute Venous ThromboEmbolism While Taking Antiplatelets
Acronym: BAT-VTE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20PH285
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Venous Thromboembolic Disease
Keywords: deep venous thrombosis; pulmonary embolism; anticoagulant; antiplatelet; Venous Thromboembolism; Direct oral anticoagulants; major adverse ischemic cardiovascular and cerebrovascular event; secondary prevention
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strategy of full-dose anticoagulant therapy alone (AC) (Experimental): The experimental group receiving full-dose anticoagulant therapy alone (AC).
  Anticoagulant (AC) therapy :at the investigator's discretion in accordance with international recommendations for the management of DVT/PE Antiplatelet therapy will be stopped.
  Interventions: Drug: Full-dose anticoagulant therapy (AC)
- strategy of combined full-dose anticoagulant and antiplatelet therapies (AC+AP) (Active Comparator): The control group receiving the standard of care: Antiplatelet therapy will be combined to full-dose anticoagulant therapy.
  Anticoagulant (AC) therapy :at the investigator's discretion in accordance with international recommendations for the management of DVT/PE
  Antiplatelet (AP) therapy : Aspirin or Clopidogrel
  Interventions: Drug: Full-dose anticoagulant therapy (AC); Drug: Antiplatelet therapy (AP)

INTERVENTIONS:
Drug: Full-dose anticoagulant therapy (AC) — Anticoagulant (AC) therapy: at the investigator's discretion in accordance with international recommendations for the management of DVT/PE
Drug: Antiplatelet therapy (AP) — Aspirin (at a daily dose ≤100 mg) or Clopidogrel (at a daily dose ≤75mg)
  Arms: strategy of combined full-dose anticoagulant and antiplatelet therapies (AC+AP)

SUMMARY:
Venous thromboembolism (VTE) and atherosclerotic cardiovascular disease share common risk factors and frequently coexist in the same patients.

Their management requires use of antithrombotic agents: anticoagulant therapy (AC) for secondary prevention of VTE recurrence, antiplatelet (AP) for secondary prevention of major adverse ischemic cardiovascular and cerebrovascular event (MACCE) in patients with atherosclerotic cardiovascular disease (coronary artery disease, atherosclerotic cerebrovascular disease, lower extremity peripheral arterial disease).

Side effects of antithrombotic drugs are the 1st cause of emergency admission and hospitalization for an adverse drug reaction (mainly bleeding), and the combination of AC with AP strongly increases this risk.

DETAILED DESCRIPTION:
Up to one third of VTE patients receive concomitant AP therapy, with conflicting results on patient outcomes. Concomitant therapy (AC+AP) has been associated with a higher risk of bleeding (up to 3-fold) when aspirin was associated with vitamin-K antagonist (VKA) in a multicenter cohort study, or with direct oral anticoagulants (DOACs) for acute VTE in a post-hoc subgroup analysis. Conversely, patients with acute VTE in whom clinicians decided to maintain AC+AP were found to have an increased risk of MACCE without any higher risk of bleeding, in a multicenter registry. However, in most cases, the type (aspirin or another) and indication (primary versus secondary prevention) of AP was unknown, as was the duration of the combination AC+AP, and therefore these observational results may be confounded. Therefore, there is persistent equipoise regarding the benefit/risk of combining an antiplatelet therapy with anticoagulation in patients undergoing treatment for VTE, when there is a prior history of atherosclerotic cardiovascular disease. This may explain why clinical practice varies widely.

Considering the conflicting data about the risk of bleeding in patients on AP therapy for secondary prevention, who need to start full-dose anticoagulant therapy for acute VTE, a randomized trial comparing the two strategies, in patients with acute VTE and with history of stable atherosclerotic cardiovascular disease is needed and justified.

The investigators hypothesize that a strategy based on the prescription of a full-dose AC therapy alone will decrease the risk of bleeding, when compared to the the strategy of combined AP and full-dose AC therapies, and that this strategy will translate in a positive net clinical benefit (a composite of clinically relevant bleeding, recurrent venous thromboembolism, and major adverse ischemic cardiovascular and cerebrovascular events).

ELIGIBILITY:
Inclusion criteria

* Signed informed consent
* Patients with acute objectively confirmed symptomatic proximal deep-vein thrombosis (DVT) or pulmonary embolism (PE) (with or without deep-vein thrombosis). Proximal deep-vein thrombosis is defined as thrombosis involving at least the popliteal vein or a more proximal vein of the lower limb.
* Indication of full-dose anticoagulant therapy for at least 3 months.
* Prescription of antiplatelet therapy for secondary prevention of atherosclerotic cardiovascular diseases, at the time of VTE diagnosis
* Life expectancy more than 3 months
* Social security affiliation

Exclusion Criteria:

* Unable to give informed consent
* Active bleeding or a high risk of bleeding contraindicating anticoagulant treatment; a systolic blood pressure of more than 180 mm Hg or a diastolic blood pressure of more than 110 mm Hg
* Anticoagulation for more than 5 days prior to randomization
* Active pregnancy or expected pregnancy or no effective contraception
* Isolated distal deep vein thrombosis
* Antiplatelet therapy prescribed for primary prevention of cardiovascular disease
* Indication to maintain a dual-antiplatelet therapy.
* Triple positive antiphospholipid syndrome, with arterial thrombosis
* Major cardiovascular and cerebrovascular event in the past 12 months for acute coronary syndrome, and in the past 6 months for cerebrovascular diseases and peripheral arterial diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant bleeding | end of the full-dose treatment period, up to 12 months
  Clinically relevant bleeding is composite of major bleeding events and clinically relevant non-major bleeding events).

SECONDARY OUTCOMES:
Net clinical benefit | end of the full-dose AC treatment period, up to 12 months
  Net clinical benefit is defined by the composite of clinically relevant bleeding, recurrent venous thromboembolism, and major adverse ischemic cardiovascular and cerebrovascular events
Clinically relevant non-major bleeding | end of the full-dose treatment period, up to 12 months
Major bleeding events | end of the full-dose treatment period, up to 12 months
recurrent venous thromboembolism | end of the full-dose treatment period, up to 12 months
  proximal deep venous thromboembolism and/or pulmonary embolism symptomatic or incidental, and including fatal-PE
arterial events | end of the full-dose treatment period, up to 12 months
  major adverse cardiovascular and cerebrovascular events (nonfatal ischemic stroke, nonfatal myocardial infarction, acute lower limb ischemia, lower limb amputation or revascularization for vascular causes, cardiovascular deaths),
venous thromboembolism (VTE) sequels | end of the full-dose treatment period, up to 12 months
  post-thrombotic syndrome (defined as a Villalta score up to 4) and post-PE syndrome (defined as the combination of a persistant dyspnea with a NYHA (New York Heart Association) scale more than I with residual vascular obstruction on lung scan

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BERTOLETTI, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (28):
- France (28):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHRU Brest - Hôpital la Cavale Blanche, Brest
  - Clinique du Parc - Castelnau-le -lez, Castelnau-le-Lez
  - CHU Clermont-Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CH le Corbusier - Firminy, Firminy
  - CHU Grenoble - Hôpital la Tronche, Grenoble
  - CH Le Puy - Hôpital Emile Roux, Le Puy-en-Velay
  - CHU Limoges, Limoges
  - HCL - Hôpital Edouard Herriot, Lyon
  - HCL - Lyon Sud, Lyon
  - APHM - Hôpital la Timone, Marseille
  - CH du Forez - Montbrison, Montbrison
  - CHU Montpellier, Montpellier
  - CHU Nancy - Hôpitaux de Brabois, Nancy
  - CHU Nantes - Hôpital Hôtel-Dieu, Nantes
  - CHU de Nice - Hôpital Pasteur, Nice
  - APHP - Hôpital Bicêtre, Paris
  - APHP - Hôpital Européen Georges Pompidou HEGP, Paris
  - APHP - Hôpital Louis Mourier, Paris
  - CHU Rouen, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CH Toulon - Hôpital Sainte Musse, Toulon
  - CHU Toulouse - Hôpital de Rangueil, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No